CLINICAL TRIAL: NCT01725555
Title: A Randomized, Open-label, Phase I, Crossover Study to Assess the Effect of Food on the Bioavailability of AXL1717, in Patients With Advanced Malignant Tumors
Brief Title: A Study to Assess the Effect of Food on the Bioavailability of the IGF-1R Inhibitor AXL1717 in Patients With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axelar AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AXL010
Record Dates: First submitted 2012-10-26; First posted 2012-11-14 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Solid Tumors; Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted treatment (Experimental)
  Interventions: Drug: Fasted treatment: AXL1717; Drug: Fed treatment: AXL1717
- Fed treatment (Experimental)
  Interventions: Drug: Fasted treatment: AXL1717; Drug: Fed treatment: AXL1717

INTERVENTIONS:
Drug: Fasted treatment: AXL1717
Drug: Fed treatment: AXL1717

SUMMARY:
This is a prospective, randomized, open-label, Phase I, crossover study to assess the effect of food on the bioavailability of AXL1717 including patients with advanced malignant tumors

DETAILED DESCRIPTION:
This is a randomized, crossover, open label, phase I study to assess the effect of food on the bioavailability of AXL1717 in advanced cancer patients.

A single, oral dose of AXL1717 is to be administered to patients on each of two occasions that are 7-day apart, in random order: after an overnight fast (fasted treatment) and with a high-fat or moderate-fat breakfast (fed treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Be informed of the nature of the study and have provided written informed consent
2. At least 18 years of age
3. Histologically confirmed diagnosis of advanced solid or hematological malignancy not amenable to standard treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 after optimization of analgesics
5. Life expectancy ≥ 3 months
6. Hematology values: blood leukocyte count ≥ 3.0 x 109/L, blood absolute neutrophil count ≥ 1.5 x 109/L, blood platelet count ≥ 100 x109/L, hemoglobin ≥ 100 g/L (transfusions are allowed)
7. Clinical chemistry values: plasma total bilirubin level ≤ 1.5 times the upper limit of the "normal" range (ULN; i.e. reference), plasma AST or ALT ≤ 1.5 x ULN (≤5 times if liver metastases have been documented) and plasma creatinine ≤ 1.5 x ULN
8. 12-lead ECG with normal tracings; or changes that are not clinically significant and do not require medical intervention

Exclusion Criteria:

1. Ongoing infection or other major recent or ongoing disease that, according to the Investigator, poses an unacceptable risk to the patient
2. Known primary or secondary central nervous system malignancy. (Patients with symptoms suggestive of possible CNS metastasis such as headache, dizziness or focal neurological deficits should undergo CT or MRI of the brain to rule out CNS metastasis. Patients who do not have CNS symptoms do not need a CT or MRI of the brain.)
3. Grade 3 or higher constipation within the past 28 days or grade 2 constipation within the past 14 days before randomization. (Patients with grade 2 constipation within the past 14 days could be re-screened if constipation decreases to ≤ grade 1 with optimal management of constipation.)
4. Impairment of gastrointestinal (GI) function, GI cancer or GI disease that may significantly alter the absorption of AXL1717
5. Coexisting uncontrolled medical condition, including active cardiac disease (such as unstable angina, myocardial infarction within 6 months, or New York Heart Association Class III/IV congestive heart failure), or significant dementia
6. Hepatic impairment as indicated by abnormalities of transaminases and/or alkaline phosphatase (AST and/or ALT > 1.5 × upper limit of normal concomitant with alkaline phosphatase > 2.5 × upper limit of normal, ≤5 times if liver metastases have been documented)
7. Major surgical procedure within 4 weeks prior to randomization
8. Use of potent inhibitors of CYP2C9 (e.g. Fluconazole) from 3 weeks prior to first administration of investigational product
9. Women of child bearing potential (WOCBP) who do not consent to using acceptable methods of contraception (i.e. two of the following - oral contraception, barrier contraception, intrauterine device). For purposes of this study, WOCBP include any female who has experienced menarche, who has not undergone tubal ligation, and who is not postmenopausal. Post menopause is defined as: amenorrhea ≥ 12 consecutive months without another cause.
10. Women who are breast-feeding or have a positive pregnancy test at screening
11. Current participation in any other investigational clinical trial or any administration of an investigational agent within 4 weeks of study drug administration or 10 half-lives of the investigational agent, whichever is longer. Patients with unresolved investigational treatment-related AEs may not participate.
12. Known or suspected hypersensitivity to AXL1717
13. Lack of suitability for participation in the trial, for any reason, as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Single dose AXL1717 serum pharmacokinetic profile under fasting versus fed condition in each patient | several samples within 24 hours

SECONDARY OUTCOMES:
Safety of AXL1717 through adverse event reporting | Up to 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Simon Ekman, M.D., Ph.D., Principal Investigator — Uppsala University Hospital, Sweden
Locations (1):
- KFUE, Uppsala, Sweden